CLINICAL TRIAL: NCT03301207
Title: A Drug-Drug Interaction Study to Evaluate the Effect of Ibrutinib on the Pharmacokinetics of Oral Contraceptives, CYP2B6, and CYP3A4 Substrates in Female Subjects With B Cell Malignancy
Brief Title: A Study to Evaluate the Effect of Ibrutinib on the Pharmacokinetics of Oral Contraceptives, CYP2B6, and CYP3A4 Substrates in Female Participants With B Cell Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108347; 2017-000496-84 (EudraCT Number); 54179060CLL1017 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Levonorgestrel; Bupropion; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib + Oral Contraceptives + Probe Drugs (CYP) (Experimental): Pre-treatment Phase: Participants will receive a single dose of oral contraceptive (OC) consisting of ethinylestradiol (EE) 30 microgram (mcg) and levonorgestrel (LN) 150 mcg on Study Day 1, and probe drugs (CYP) consisting of bupropion 75 milligram (mg) and midazolam 2 mg on Study Day 3, followed by a washout period from Study Days 4 to 7. Treatment Phase: Participants will receive ibrutinib 560 mg (4*140 mg capsules) once daily (QD) on Days 8 to 26 along with midazolam 2 mg once orally on Study Day 8 (Cycle 1 Day 1), OC once orally on Study Day 22 (Cycle 1 Day 15; EE and LN), and bupropion 75 mg and midazolam 2 mg once orally on Study Day 24 (Cycle 1 Day 17). From Study Day 27 (Cycle 1 Day 20) and onwards participants will continue oral treatment with ibrutinib 420 mg (3*140 mg capsules) or 560 mg QD (depending on the subtype of B-cell malignancy) up to the end of Cycle 6 (each cycle will consist of 28 days).
  Interventions: Drug: Ibrutinib; Drug: OC: Ethinylestradiol (EE) 30 mcg and Levonorgestrel (LN) 150 mcg; Drug: Bupropion; Drug: Midazolam

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib capsule (at dose of 420 or 560 mg) will be taken orally QD.
  Other Names: Imbruvica
Drug: OC: Ethinylestradiol (EE) 30 mcg and Levonorgestrel (LN) 150 mcg — Single dose of oral contraceptives (OC) (1 tablet containing 30 mcg EE and 150 mcg LN) will be taken orally on Study Days 1 and 22.
  Other Names: Microgynon 30
Drug: Bupropion — Bupropion 75 mg tablet as a part of CYP cocktail will be taken on Study Days 3 and 24.
Drug: Midazolam — Midazolam 2 mg (1 milliliter [mL]) oral solution will be taken on Study Days 3 and 24 (as a part of CYP cocktail) and on Study Day 8 (alone).

SUMMARY:
The main purpose of this study is to evaluate the effects of repeat dosing of ibrutinib on the single-dose pharmacokinetics (PK) of oral contraceptives (OC - ethinylestradiol [EE] and levonorgestrel [LN]), the cytochrome P450 (CYP)2B6 probe bupropion and the CYP3A4 probe midazolam; and to evaluate the effects of single-dose ibrutinib on the single-dose PK of the CYP3A4 probe midazolam in female participants with B cell malignancy.

DETAILED DESCRIPTION:
This is a multicenter study of ibrutinib (first-in-class, potent, covalently-binding inhibitor of Bruton's tyrosine kinase [BTK]) in female participants with B cell malignancy. The study consists of 3 phases: Screening Phase (up to 28 days), 7-day Pretreatment Phase (Days 1 to 7), Treatment Phase including PK assessment period (Days 8 to 26) and a Follow-up Phase (Day 27 to end of Cycle 6). The study procedures includes electrocardiogram (ECG), vital signs, blood samples withdrawal to evaluate PK and safety. The Antitumor activity will be assessed by means of computed tomography (CT) imaging and positron emission tomography (PET) scans. No formal statistical hypothesis will be tested. This is an estimation study designed to determine if an increase or decrease in exposure to OC or probe drugs occurs in the presence of ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL), or Waldenstrom's macroglobulinemia (WM)

  1. Participants with MCL must have relapsed or refractory disease after at least 1 prior line of systemic therapy
  2. Participants with MZL must have failed an anti-cluster of differentiation (CD)20 monoclonal antibody-based therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Adequate hematologic, hepatic, and renal functions
* Before the first dose of oral contraceptive (OC), a woman must be either:

  1. Not of childbearing potential: postmenopausal (greater than [>]45 years of age with amenorrhea for at least 12 months and a serum follicle stimulating hormone level >40 international unit per Liter [IU/L] or milli international unit per milli Liter [mIU/mL]); permanently sterilized
  2. Of childbearing potential and practicing a highly effective non-hormonal method of birth control
* Women of childbearing potential must have a negative serum (Beta-human chorionic gonadotropin [Beta-hCG]) or urine pregnancy test at screening

Exclusion Criteria:

* Major surgery planned within 2 weeks of the first dose of ibrutinib or during study participation up to Cycle 2 Day 1
* History of other malignancies, except:

  1. Malignancy treated with curative intent and with no known active disease present for greater than or equal to (>=)3 years before the first dose of ibrutinib and felt to be at low risk for recurrence by treating physician
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated in-situ cancer without evidence of disease
* History of breast or endometrial cancer
* Prior treatment/exposure with ibrutinib or other Bruton's tyrosine kinase (BTK) inhibitor
* Requires ongoing anticoagulation treatment with warfarin or equivalent vitamin K antagonists (for example, phenprocoumon)
* Requires therapies that must be discontinued or substituted 7 days prior to Study Day 1, or must be temporally interrupted during the course of the study, including the following:

  1. Medications known to induce or inhibit drug metabolizing enzymes (CYP3A4 and CYP2B6)
  2. Medication which are not allowed to be used in combination with EE, LN, bupropion, or midazolam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Ethinylestradiol (EE) and Levonorgestrel (LN) When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 1 and 22: predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, and 72 hours (h) post-dose
  The Cmax is the maximum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) of Bupropion and 4-Hydroxybupropion When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 3 and 24: predose, 0.5, 1, 2, 3, 4, 6, 10, 24, 34, 48, 58 h post-dose
  The Cmax is the maximum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Repeat Doses of Ibrutinib | Day 3: predose, 15 minutes (min), and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 24: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 24 h post-dose
  The Cmax is the maximum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Single Dose of Ibrutinib | Day 3: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 8: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 12 h post-dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of EE and LN When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 1 and 22: predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, and 72 h post-dose
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of Bupropion and 4-Hydroxybupropion When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 3 and 24: predose, 0.5, 1, 2, 3, 4, 6, 10, 24, 34, 48, 58 h post-dose
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Repeat Doses of Ibrutinib | Day 3: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 24: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 24 h post-dose
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Single Dose of Ibrutinib | Day 3: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 8: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 12 h post-dose
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of EE and LN When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 1 and 22: predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, and 72 h post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Bupropion and 4-Hydroxybupropion When Co-administered With Repeat Doses of Ibrutinib Compared to Administration Alone | Days 3 and 24: predose, 0.5, 1, 2, 3, 4, 6, 10, 24, 34, 48, 58 h post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Repeat Doses of Ibrutinib | Day 3: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 24: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 24 h post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Midazolam and 1-Hydroxymidazolam When Co-Administered With Single Dose of Ibrutinib | Day 3: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10,12, and 24 h post-dose; Day 8: predose, 15 min, and 0.5,1,2,3,4,5,6,8,10, and 12 h post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Plasma Concentration of Ibrutinib and its Metabolite PCI-45227 | Predose, 1, 2, 4, and 6 h post-dose on Days 8, 22, and 24
  Plasma concentrations of Ibrutinib and its Metabolite PCI-45227 will be measured.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Screening up to end of the 6 month treatment or 30 days after the last dose of study drug for Participants discontinuing treatment before 6 months
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants With Laboratory Abnormalities as a Measure of Safety and Tolerability | Screening, Days 8 and 36, and End of Treatment (approximately 7 months)
  Blood samples for serum chemistry and hematology will be collected at predefined time points for clinical laboratory testing.
Number of Participants With Electrocardiogram (ECG) Abnormalities Findings as a Measure of Safety and Tolerability | Screening and End of Treatment (approximately 7 months)
  Triplicate ECG will be performed at screening and a single time point ECG will be performed at end of treatment visit.
Number of Participants With Vital Sign Abnormalities as a Measure of Safety and Tolerability | Screening, Days 8 and 36, and End of Treatment (approximately 7 months)
  Vital signs includes Temperature, Heart Rate, Respiratory Rate and Blood Pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Spain (2):
  - Hosp. Univ. Fund. Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona

REFERENCES:
- [Derived] de Jong J, Mitselos A, Jurczak W, Cordoba R, Panizo C, Wrobel T, Dlugosz-Danecka M, Jiao J, Sukbuntherng J, Ouellet D, Hellemans P. Ibrutinib does not have clinically relevant interactions with oral contraceptives or substrates of CYP3A and CYP2B6. Pharmacol Res Perspect. 2020 Oct;8(5):e00649. doi: 10.1002/prp2.649. PMID 32945596
- See also: A Drug-Drug Interaction Study to Evaluate the Effect of Ibrutinib on the Pharmacokinetics of Oral Contraceptives, CYP2B6, and CYP3A4 Substrates in Female Subjects with B Cell Malignancy — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108347&attachmentIdentifier=81191578-48db-427d-b269-9351a0c2e39a&fileName=CR108347_CSR_Synopsis.pdf&versionIdentifier=